CLINICAL TRIAL: NCT05557487
Title: Taiwan Real-world Low-dose Computed Tomography Screening behavIor and Outcome Research for High Risk Subjects Based on Health Promotion Administration-part A: Questionnaire Survey -Part B: LDCT Screening Outcome and Management
Brief Title: Taiwan Real-world LDCT Screening Behavior and Outcome Research for High Risk Subjects Based on Health Promotion Administration
Acronym: TRIO
Status: Recruiting | Type: Observational
Sponsor: Gee-Chen Chang (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor-Investigator, Gee-Chen Chang, Chung Shan Medical University, Chung Shan Medical University
Organization: Chung Shan Medical University (Other)
Other Study IDs: CS1-22111
Record Dates: First submitted 2022-09-23; First posted 2022-09-28 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Lung Cancer; High-Risk Cancer; Smoking; Pollution; Exposure; Family Relations
Keywords: Lung cancer; Low-dose computed tomography; Real world data; Lung cancer family history; Air pollution; Smoking; Lung cancer risk questionnaire
MeSH Terms: conditions — Lung Neoplasms; Smoking | interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples, urine samples, lung tissue samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Previous heavy smokers: Age 40 to 80 years who have at least a 20-pack-year smoking history with successful smoking cessation history (stopping smoking for more than 6 months), but less than 15 years
  Interventions: Diagnostic Test: Low dose computed tomography
- First degree relatives of lung cancer patients: First-degree relatives of lung cancer patients
  1. aged more than 40 years
  2. age less than 40 years old, but older than the age at diagnosis of the youngest lung cancer proband in the family
  Interventions: Diagnostic Test: Low dose computed tomography
- With other high-risk occupational or environmental factors: Age 40 to 80 years, meet one or more of the following criteria.
  1. air-pollution exposed occupations (such as traffic policeman, street cleaners….) for at least 10 years
  2. cooking index ≥ 110, defined as 2/7 * days cooking by pan frying, stir frying, or deep frying in one week * years cooking.
  3. cooking without using ventilation for more than 20 years
  4. history of pulmonary tuberculosis and complete anti-tuberculosis treatment with interval more than 5 years before this study
  Interventions: Diagnostic Test: Low dose computed tomography

INTERVENTIONS:
Diagnostic Test: Low dose computed tomography — 1. Participants belonging to modified Lung RADS category 1 and 2 at baseline screening will undergo the LDCT next year after the discussion with the physicians in charge.
  2. Participants with nodules belonging to modified Lung RADS category 3 and 4, growing nodules, or new nodules found on follow-up LDCT scans will undergo repeat CT every 3 to 6 months or be referred for diagnostic workup depending on the size and characteristics of the nodules as the regular clinical practice.
  3. Volume doubling time (VDT) will be performed in the special groups with Lung RADS category 3 or 4, but the nodules with solid components ≧ 6mm and < 9mm. A repeat LDCT scan will be performed around 3 months after the baseline screening.
  4. Check total bilirubin, urinary heavy metals,CRP, serum tumor marker, including CEA, alpha-fetal protein, etc.
  5. Check pulmonary function test.

SUMMARY:
Lung cancer is the leading cause of mortality in the world, and also in Taiwan.Despite the researches and availability in new therapies, it causes the highest mortality and is one of the most preventable cancers as well. Smoking is the most common cause of lung cancer worldwide. Compared to lung cancer in smokers, lung cancer in never-smokers is associated with East Asian ethnicity, female sex, and adenocarcinoma histology. This unique risk group is likely to have distinct molecular drivers, especially EGFR, ALK, and ROS1 mutations.In National Taiwan Cancer Registry data, more than half (53%) of all newly diagnosed lung cancer patients and 93% of female patients are lifelong never-smokers. This scenario is common in East Asia. It is essential to develop a different strategy for screening lung cancer patients with other high-risk profiles. Several risk factors have been identified in never-smoking lung cancer and one of the most important factor is a lung cancer family history (LCFH) in a first-degree relative. Other high-risk occupational or environmental factors include air-pollution exposed occupations (such as traffic policeman and street cleaners) for at least 10 years, cooking index ≥ 110, defined as 2/7 * days cooking by pan frying, stir frying, or deep frying in one week * years cooking, cooking without using ventilation, passive smoke exposure, and history of pulmonary tuberculosis or chronic obstructive pulmonary disorders.

As described above, three high risk groups are interested in this study, the previous heavy smokers (group 1); those who has family history (group 2) and those who have high risk occupation or environment factors (group 3). From the published researches, we assume the detection rate to be 1.1% for group 1 based on NLST results16, 2.6% for group 2 (395 out of 12,011 subjects in TALENT), and we assume the detection Group 3 to be 1% after consulting board-certified senior specialists in this field.

This is a prospective, multi-center, single arm study in Taiwan of subjects who are eligible to receive LDCT screening based on recommendation of Health Promotion Administration of Taiwan.

The primary objective of TRIO part A is the LDCT screening acceptance rate of high lung cancer risk subjects.

The primary objective of TRIO part B is the exact lung cancer detection rates in these three groups.

Other secondary objectives are also included.

ELIGIBILITY:
Inclusion Criteria:

Group 1: Previous heavy smokers Age 50 to 80 years, meet both criteria in the followings.

1. Cigarette smoking of at least 20 pack-years
2. With successful smoking cessation history (stopping smoking for more than 6 months), but less than 15 years

Group 2: First-degree relatives of lung cancer patients

1. aged more than 50 years
2. age less than 50 years old, but older than the age at diagnosis of the youngest lung cancer proband in the family

Group 3: With other high-risk occupational or environmental factors Age 50 to 80 years, meet one or more of the following criteria.

1. air-pollution exposed occupations (such as traffic policemen, and street cleaners….) for at least 10 years
2. cooking index ≥ 110, defined as 2/7 * days cooking by pan frying, stir-frying, or deep frying in one week * years cooking.
3. cooking without using ventilation for more than 20 years
4. history of pulmonary tuberculosis and complete anti-tuberculosis treatment with intervals more than 5 years before this study

Exclusion Criteria:

1. previous history of lung cancer
2. another malignancy except for cervical carcinoma in situ or non-melanomatous carcinoma of the skin within 5 years
3. an inability to tolerate transthoracic procedures or thoracotomy
4. chest CT examination was performed within 18 months
5. hemoptysis of unknown etiology within one month
6. body weight loss of more than 6 kg within one year without an evident cause
7. a known pregnancy
8. Not capable of understanding or responding to the written questionnaire even through the help from the study team

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: High risk population for lung cancer
Sampling Method: Non-Probability Sample
Enrollment: 6618 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
The rate of willingness and completeness of LDCT screening after the detailed questionnaire survey for the eligible participants. | 2 years
  1. Eligible participants must meet the inclusion and exclusion criteria of this study
  2. Only the one who completes the detailed questionnaire survey is counted.
To investigate overall lung cancer detection rate of high lung cancer risk individuals | 2 years
  Cytological or Pathological proof of lung cancer to investigate the overall lung cancer detection rate

CONTACTS AND LOCATIONS:
Locations (7):
- Taiwan (7):
  - Chung Shan Medical University, Taichung, Taiwan
  - National Taiwan University Hospital Hsin-Chu Branch, Hsinchu
  - Hualien Tzu Chi Hospital, Hualien City
  - E-Da Hospital, Kaohsiung City
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Ministry of Health and Welfare Shuang-Ho Hospital, New Taipei City
  - National Taiwan University Hospital, Taipei

REFERENCES:
- [Background] Torre LA, Bray F, Siegel RL, Ferlay J, Lortet-Tieulent J, Jemal A. Global cancer statistics, 2012. CA Cancer J Clin. 2015 Mar;65(2):87-108. doi: 10.3322/caac.21262. Epub 2015 Feb 4. PMID 25651787
- [Background] National Lung Screening Trial Research Team; Church TR, Black WC, Aberle DR, Berg CD, Clingan KL, Duan F, Fagerstrom RM, Gareen IF, Gierada DS, Jones GC, Mahon I, Marcus PM, Sicks JD, Jain A, Baum S. Results of initial low-dose computed tomographic screening for lung cancer. N Engl J Med. 2013 May 23;368(21):1980-91. doi: 10.1056/NEJMoa1209120. PMID 23697514
- [Background] Patz EF Jr, Pinsky P, Gatsonis C, Sicks JD, Kramer BS, Tammemagi MC, Chiles C, Black WC, Aberle DR; NLST Overdiagnosis Manuscript Writing Team. Overdiagnosis in low-dose computed tomography screening for lung cancer. JAMA Intern Med. 2014 Feb 1;174(2):269-74. doi: 10.1001/jamainternmed.2013.12738. PMID 24322569
- [Background] US Preventive Services Task Force; Krist AH, Davidson KW, Mangione CM, Barry MJ, Cabana M, Caughey AB, Davis EM, Donahue KE, Doubeni CA, Kubik M, Landefeld CS, Li L, Ogedegbe G, Owens DK, Pbert L, Silverstein M, Stevermer J, Tseng CW, Wong JB. Screening for Lung Cancer: US Preventive Services Task Force Recommendation Statement. JAMA. 2021 Mar 9;325(10):962-970. doi: 10.1001/jama.2021.1117. PMID 33687470
- [Background] Kim H, Kim HY, Goo JM, Kim Y. Lung Cancer CT Screening and Lung-RADS in a Tuberculosis-endemic Country: The Korean Lung Cancer Screening Project (K-LUCAS). Radiology. 2020 Jul;296(1):181-188. doi: 10.1148/radiol.2020192283. Epub 2020 Apr 14. PMID 32286195
- [Background] de Koning HJ, van der Aalst CM, de Jong PA, Scholten ET, Nackaerts K, Heuvelmans MA, Lammers JJ, Weenink C, Yousaf-Khan U, Horeweg N, van 't Westeinde S, Prokop M, Mali WP, Mohamed Hoesein FAA, van Ooijen PMA, Aerts JGJV, den Bakker MA, Thunnissen E, Verschakelen J, Vliegenthart R, Walter JE, Ten Haaf K, Groen HJM, Oudkerk M. Reduced Lung-Cancer Mortality with Volume CT Screening in a Randomized Trial. N Engl J Med. 2020 Feb 6;382(6):503-513. doi: 10.1056/NEJMoa1911793. Epub 2020 Jan 29. PMID 31995683